CLINICAL TRIAL: NCT00835861
Title: Pilot Study of Metformin vs. Insulin in Pregnant Overt Diabetics (MIPOD)
Brief Title: Effectiveness of Metformin Compared to Insulin in Pregnant Women With Mild Preexisting or Early Gestational Diabetes
Acronym: MIPOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: WakeMed Health and Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNC08-0898
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2014-04

CONDITIONS: Non Insulin Dependent Diabetes; Pregnancy
Keywords: Non Insulin Dependent Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Insulin; Insulin, Isophane; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Women who enter pregnancy with a diagnosis of non insulin dependent/Type 2 Diabetes that is controlled with diet or an oral hypoglycemic agent, and women who demonstrate abnormal glucose tolerance prior to 20 weeks of gestation by abnormal 3 hour glucose challenge testing will be offered study participation. After informed consent, they will be randomized 1:1 to either the Metformin or Insulin group.
  Interventions: Drug: Metformin
- Insulin (Active Comparator): Women who enter pregnancy with a diagnosis of non insulin dependent/Type 2 Diabetes that is controlled with diet or an oral hypoglycemic agent, and women who demonstrate abnormal glucose tolerance prior to 20 weeks of gestation by abnormal 3 hour glucose challenge testing will be offered study participation. After informed consent, they will be randomized 1:1 to either the Metformin or Insulin group.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — Women randomized to the Experimental arm will receive standard diet and glucose self-monitoring education. They will be initiated on Metformin 500 BID if they were medication naïve, or will be continued on their current dosage of Metformin if they were taking it prior to pregnancy. At each clinic visit fasting and one hour post prandial glucose values will be reviewed, and dosage will be titrated to a maximum of 2250mg/day to achieve target glycemic control. If glycemic control can not be achieved with Metformin as a single agent insulin will be added.
  Other Names: Glucophage
  Arms: Metformin
Drug: Insulin — Women randomized to the Insulin group will receive standard diet and glycemic monitoring education. They will be initiated on weight based Regular and NPH insulin at a total dosage of 0.7units/kg in the first trimester or 0.8units/kg in the second trimester divided as 2/3 of the total dosage (with 2/3 given as NPH and 1/3 given as Regular) administered before breakfast and 1/3 of the total dosage (with 1/2 given as NPH and 1/2 given as Regular)administered with dinner. At each clinic visit fasting and one hour post prandial glucose values will be reviewed, and dosage will be titrated to achieve optimal glycemic control with fasting values <90 and one hour post prandial values <130.
  Other Names: Regular Insulin; Novolin R; Humulin R; NPH Insulin; Novolin N; Humulin N
  Arms: Insulin

SUMMARY:
Many women come into pregnancy with diabetes that is controlled with either Metformin or diet control; however, the current standard of care for the treatment of preexisting diabetes in pregnancy is insulin. Metformin is widely used in the non-pregnant population for glycemic control, and has been used in pregnancy for other indications without adverse maternal or fetal outcomes. What remains unproven is the ability of Metformin to adequately control glucose in women during pregnancy.

Our goal is to randomize 100 women who enter pregnancy with diabetes that is controlled by either diet or an oral agent and women who are found to have an abnormal glucose challenge test at less than 20 weeks to either standard treatment with weight based Regular and neutral protamine Hagedorn (NPH) insulin or Metformin. Our hypothesis is that Metformin will provide glycemic control that is equivalent to insulin in these women.

ELIGIBILITY:
Inclusion Criteria:

* Receiving prenatal care at University of North Carolina (UNC), Chapel Hill Obstetric clinics and planning delivery at UNC Women's Hospital
* Diagnosis of Diabetes prior to pregnancy with use of an oral hypoglycemic agent or dietary control
* Diagnosis of early gestational diabetes prior to 20 weeks gestation via abnormal 3 hour glucose challenge testing using the national diabetes data group (NDDG)criteria
* Less than 24 weeks at study enrollment
* Singleton or twin pregnancy
* English or Spanish speaking
* Able to give informed consent

Exclusion Criteria:

* End organ complications of diabetes (retinopathy, renal insufficiency, etc.)
* Prior need for insulin for glycemic control
* History of diabetic ketoacidosis (DKA) or hyperosmolar state
* Prior adverse reaction (ie. lactic acidosis) or allergy to Metformin
* Kidney or liver disease
* Significant medical co-morbidities (lupus, cystic fibrosis, etc.) Hypertension controlled on one medication, well controlled asthma, and well controlled thyroid disease are not excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Hickman, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals Obstetric Clinics, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Hickman MA, McBride R, Boggess KA, Strauss R. Metformin compared with insulin in the treatment of pregnant women with overt diabetes: a randomized controlled trial. Am J Perinatol. 2013 Jun;30(6):483-90. doi: 10.1055/s-0032-1326994. Epub 2012 Oct 24. PMID 23096052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at two hospitals from July 2008 through March 2010 at one and from January 2009 through December 2009 at the other.
Groups:
- Metformin: Patients received standard diet and glucose self-monitoring education. Medication naive patients were initiated on Metformin 500 BID or were continued on their current dosage of Metformin if taking prior to pregnancy. Self-reported glucose values were reviewed during each clinic visit and Metformin dosage was titrated up to a maximum of 2250 mg/day as needed for glycemic control. Insulin was added to those not achieving glycemic control with Metformin alone
- Insulin: Patients received standard diet and glycemic monitoring education. They were started on weight-based Regular and neutral protamine Hagedorn (NPH) insulin at a total dosage of 0.7units/kg in the first trimester or 0.8units/kg in the second trimester divided as 2/3 of the total dosage (with 2/3 given as NPH and 1/3 given as Regular) administered before breakfast and 1/3 of the total dosage (with 1/2 given as NPH and 1/2 given as Regular) administered with dinner. Self-reported glucose values were reviewed during each clinic visit and insulin dosage was titrated to achieve optimal glycemic control with fasting values <90 and one hour post prandial values <130.
Period: Overall Study
Arm/Group | Metformin | Insulin
Started | 15 | 16
Completed | 14 | 14
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Three women who never received the allocated treatment were excluded from the analysis.
Groups:
- Insulin: Patients received standard diet and glycemic monitoring education. They were started on weight-based Regular and NPH insulin at a total dosage of 0.7units/kg in the first trimester or 0.8units/kg in the second trimester divided as 2/3 of the total dosage (with 2/3 given as NPH and 1/3 given as Regular) administered before breakfast and 1/3 of the total dosage (with 1/2 given as NPH and 1/2 given as Regular) administered with dinner. Self-reported glucose values were reviewed during each clinic visit and insulin dosage was titrated to achieve optimal glycemic control with fasting values <90 and one hour post prandial values <130.
- Total: Total of all reporting groups
Arm/Group | Metformin | Insulin | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (2.6) | 29.7 (4.1) | 32.7 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Measurements
Description: Patients self monitored glucose measures throughout pregnancy to aid glycemic control. Fasting morning measures and postprandial measures were taken at 1 hour after breakfast, lunch, and dinner.
Time Frame: Daily fasting and 1-hr post prandial measures were taken from time of enrollment until delivery
Population: For 1 infant in each group, the initial neonatal glucose value was missing.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Metformin: Standard diet and glucose self-monitoring education. Initiated on Metformin 500 BID if medication naïve, or continued on their current dosage of Metformin if taking it prior to pregnancy. Dosage titrated to a maximum of 2250 mg/day based on review of self-reported fasting and post prandial glucose values during visits. .NPH Insulin treatment added for those unable to achieve glycemic control with Metformin alone.
- Insulin: Standard diet and glycemic monitoring education. Initiated on weight-based Regular and NPH insulin at a total dosage of 0.7units/kg in the first trimester or 0.8units/kg in the second trimester divided as 2/3 of the total dosage (with 2/3 given as NPH and 1/3 given as Regular) administered before breakfast and 1/3 of the total dosage (with 1/2 given as NPH and 1/2 given as Regular) administered with dinner. Dosage titrated during visits to achieve optimal glycemic control with fasting values <90 mg/dL and 1-hr post prandial values < 130 mg/dL.
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
mg/dL
  Fasting throughout enrollment | 97.38 [92 to 101] | 95.04 [86 to 115]
  Fasting 18-20 weeks | 97.00 [93 to 100] | 92.38 [89 to 116]
  Fasting 28-30 weeks | 92.43 [90 to 98] | 90.64 [84 to 106]
  Fasting 36-38 weeks | 89.49 [82 to 96] | 85.18 [80 to 107]
  Postprandial throughout enrollment | 120.40 [115 to 129] | 128.62 [115 to 143]
  Postprandial 18-20 weeks | 118.40 [107 to 122] | 120.46 [113 to 142]
  Postprandial 28-30 weeks | 119.00 [114 to 125] | 126.45 [115 to 137]
  Postprandial 36-38 weeks | 122.59 [118 to 130] | 125.25 [112 to 138]

2. Secondary Outcome: Number of Patients With Obstetric Complications
Description: Maternal complications were stillbirths, major malformations, shoulder dystocia, or postpartum hemorrhage requiring transfusion.
Time Frame: Throughout pregnancy until hospital discharge following delivery.
Measure: Number; unit: participants
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
participants | 0 | 0

3. Secondary Outcome: Maternal Weight Gain
Time Frame: Baseline throughout pregnancy until last prenatal visit.
Measure: Median (Inter-Quartile Range); unit: kg/week
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
kg/week | 0.28 [0.11 to 0.38] | 0.30 [0.18 to 0.47]

4. Secondary Outcome: Number of Babies With Neonatal Hypoglycemia
Description: Initial neonatal glucose < 40 mg/dL
Time Frame: Time of delivery through hospital discharge
Population: For 1 infant in each group, the initial neonatal glucose value was missing.
Measure: Number; unit: Number of babies
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 13 | 13
Number of babies | 2 | 0

5. Secondary Outcome: Glycosylated Hemoglobin (HbA1c) by Pregnancy Trimester
Time Frame: 1st, 2nd, and 3rd trimester
Measure: Median (Inter-Quartile Range); unit: percentage of glycosolated hemoglobin
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
percentage of glycosolated hemoglobin
  1st trimester | 5.8 [5.4 to 6.5] | 6.2 [5.7 to 7.5]
  2nd trimester | 5.6 [5.4 to 5.8] | 5.5 [5.2 to 6.1]
  3rd trimester | 5.9 [5.5 to 6.0] | 5.6 [5.3 to 6.4]

6. Secondary Outcome: Percent of Glucose Values at or Below Fasting Goal (<95 mg/dL)
Description: NUMBER OF ASSESSMENTS OF FASTING GLUCOSE VALUES <95
Time Frame: Baseline throughout pregnancy until time of delivery
Measure: Number; unit: percent of glucose values
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
percent of glucose values
  Throughout enrollment; n=1634, 1432 | 48 [0.38 to 0.67] | 58 [0.17 to 0.81]
  18-20 weeks; n=148, 259 | 42 [0.31 to 0.57] | 64 [0.00 to 0.83]
  28-30 weeks; n=253, 201 | 64 [0.29 to 0.85] | 62 [0.23 to 1.00]
  36-38 weeks; n=115, 83 | 76 [0.54 to 0.93] | 96 [0.20 to 1.00]

7. Secondary Outcome: Percent of Glucose Values at or Below Postprandial Goal (<130 mg/dL)
Description: NUMBER OF ASSESSMENTS OF POSTPRANDIAL GLUCOSE VALUES <130
Time Frame: Baseline throughout pregnancy until time of delivery
Measure: Number; unit: percent of glucose values
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
percent of glucose values
  Throughout enrollment; n=4195, 3796 | 69 | 61
  18-20 weeks; n=368, 428 | 72 | 67
  28-30 weeks; n=652, 559 | 71 | 58
  36-38 weeks; n=272,228 | 66 | 65

8. Secondary Outcome: Number of Episodes Maternal Hypoglycemia
Description: Maternal glucose < 60 mg/dL
Time Frame: Baseline throughout pregnancy until time of delivery
Measure: Number; unit: Number of episodes
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 14 | 14
Number of episodes | 1 | 7

9. Secondary Outcome: Number of Babies With Adverse Neonatal Outcomes
Description: Resuscitation in the delivery room, preterm birth < 37 weeks, neonatal intensive care unit care, birth injury or diagnosis of neonatal complication, glucose infusion, antibiotics, or phototherapy.
Time Frame: Delivery until hospital discharge
Population: For 1 infant in the metformin group, the "adverse neonatal outcome" data was missing.
Measure: Number; unit: number of babies
Arm/Group | Metformin | Insulin
Number analyzed (Participants) | 13 | 14
number of babies | 4 | 7

ADVERSE EVENTS:
Time Frame: From July 2008 through March 2010
Arm/Group | Metformin | Insulin
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=14) | Insulin (N=14)
Intrauterine fetal demise (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — In the metformin group, one woman experienced a 13-week intrauterine fetal demise attributed to a large subchorionic hematoma noted on ultrasound at 12 weeks.

LIMITATIONS AND CAVEATS:
Unable to achieve enrollment goal before funding period expired because recruitment progressed more slowly than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No